CLINICAL TRIAL: NCT03260127
Title: Enhancement of PTSD Treatment With Computerized Executive Function Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F2459-W; IK2RX002459 (NIH)
Record Dates: First submitted 2017-08-09; First posted 2017-08-24 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; treatment; posttraumatic stress disorder; therapy; cognition; thinking; executive function; computer; training
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CEFT-CPT (Experimental): Computerized executive function training plus Cognitive Processing Therapy for PTSD
  Interventions: Behavioral: Computerized executive function training plus CPT (CEFT-CPT)
- WT-CPT (Active Comparator): Word game training plus Cognitive Processing Therapy for PTSD
  Interventions: Behavioral: Word game training plus CPT (WT-CPT)

INTERVENTIONS:
Behavioral: Computerized executive function training plus CPT (CEFT-CPT) — Participants randomized to the CEFT-CPT arm will receive 6 weeks of computerized executive function training and then 6 weeks of standard Cognitive Processing Therapy for PTSD (total of 12 sessions)
  Arms: CEFT-CPT
Behavioral: Word game training plus CPT (WT-CPT) — Participants randomized to the WT-CPT arm will receive 6 weeks of computerized word game training and then 6 weeks of standard Cognitive Processing Therapy for PTSD (total of 12 sessions)
  Arms: WT-CPT

SUMMARY:
This study focuses on helping Iraq and Afghanistan Veterans with posttraumatic stress disorder (PTSD) benefit fully from therapy by first enhancing their thinking abilities. PTSD has been associated with thinking problems, including difficulty planning/organizing, thinking flexibly, and inhibiting distracting emotional information. There is some evidence that computerized training programs are helpful for improving thinking. Therefore, this study tests whether computerized cognitive training will in fact improve individuals' thinking abilities and if this will in turn improve PTSD treatment outcomes and lead to more individuals completing treatment and showing greater improvements in emotional symptoms and quality of life than standard therapy (when paired with a word training condition).

DETAILED DESCRIPTION:
PTSD affects approximately 14% of OEF/OIF Veterans and leads to considerable personal and societal costs (e.g., increased morbidity, reduced work productivity, poorer relationships). Although cognitive behavioral therapy (CBT) is one of the most effective treatments for PTSD, a substantial portion (approximately 50%) of individuals drop out prematurely, do not respond to treatment, or relapse.

Treatment engagement is worse for OEF/OIF Veterans, who attend fewer sessions and have higher dropout rates than civilians and Veterans from other eras. One likely barrier to treatment engagement and effectiveness is the executive functioning problems present in individuals with PTSD. Executive functions (EFs) are the set of higher-level cognitive skills that organize and integrate lower-level cognitive processes in order to perform complex, goal-directed tasks. PTSD has been associated with EF deficits, including impairments in inhibitory control, working memory, and cognitive flexibly, as well as dysfunction in a network of brain regions that support EFs (e.g., prefrontal cortex [PFC], cingulate).

EFs are essential for CBT in order to engage the cognitive skills involved in treatment (e.g., self-monitoring, inhibiting distorted thoughts, and flexibly generating/evaluating alternative thoughts). This is particularly true for Cognitive Processing Therapy (CPT), a frontline CBT treatment for PTSD, which involves identifying and challenging maladaptive trauma-related thoughts to alter their impact on emotions and behavior. Thus, EF deficits may lead to reduced CPT engagement and responsivity. In fact, worse EF at baseline has been associated with poorer response to CBT in several disorders (e.g., generalized anxiety disorder, obsessive compulsive disorder, and schizophrenia). Further, a study of brain functioning during an EF task demonstrated that dysfunction in EF-related brain regions including PFC and cingulate cortex at baseline predicted nonresponse to CBT for PTSD. Directly targeting EF prior to CPT via cognitive training would strengthen executive networks and likely boost treatment effectiveness, allowing Veterans to fully engage in and benefit more from components of CPT (e.g., cognitive restructuring). Evidence suggests that computerized cognitive training improves EF and functioning in EF-related brain regions, increases mental health treatment completion rates, and goal of the proposed study is to examine whether administering computerized EF training (CEFT) immediately prior to CPT will improve executive functioning and enhance treatment adherence, completion rates, and psychological and functional outcomes in OEF/OIF Veterans with PTSD.

Objective (neuropsychological) and subjective (self- report) measures of EF will be collected to determine if CEFT enhances EF and if this in turn mediates the relationship between treatment condition and PTSD symptom improvement. Functional neuroimaging during EF tasks will also be collected at baseline to determine whether functioning within an EF network predicts treatment response, above and beyond traditional paper-and-pencil measures of EF. Veterans will be randomized to either 12 weeks of CEFT-CPT or a placebo word training condition plus CPT.

Assessments will be administered at baseline, immediately after CEFT or word training (prior to CPT), and after CPT completion. The proposed research aims to reduce barriers to treatment engagement and has potential to significantly enhance current treatments for PTSD by combining cognitive and psychotherapeutic approaches. Targeting EF directly and independently represents a logical, innovative, and empirically-informed method for augmenting existing treatments for PTSD in order to optimize outcomes. Findings from the proposed study will not only directly inform clinical practice, but also have the potential to significantly improve the quality of Veterans' lives, reduce societal costs and burden, improve access to care, and reveal ways to better match individuals with treatments they are most likely to benefit from.

ELIGIBILITY:
Inclusion Criteria:

* Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans enrolled at Veterans Affairs San Diego Healthcare System (VASDHS)
* aged 18-55
* current posttraumatic stress disorder (PTSD) diagnosis
* endorsement of cognitive complaints
* no pending medication changes
* English-speaking.

Exclusion Criteria:

* active substance use disorder in the last month
* suicidal intent or attempt within the last month
* schizophrenia, psychotic disorder and/or bipolar disorder
* dementia
* premorbid IQ < 70
* participation in other concurrent PTSD intervention studies
* previous completion of more than 4 Cognitive Processing Therapy (CPT) sessions
* history of a documented neurological disorder (e.g., Parkinson's disease, multiple sclerosis, epilepsy)
* moderate to severe traumatic brain injury (TBI) (i.e., loss of consciousness greater than 30 minutes or post-traumatic amnesia greater than 24 hours).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura D. Crocker, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Requests for access must be made in writing signed by a requestor from the United States and include an email address for delivery and an assurance that the recipient will not attempt to identify or re-identify any individual. The request should reference the publication underlying the request. Requests may be made to the Principal Investigator/lead point-of-contact for the publication. If the investigator leaves the VA San Diego Healthcare System, the requests may be sent to the Associate Chief of Staff for Research.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who were were enrolled were randomly assigned to groups.
Period: Overall Study
Arm/Group | CEFT-CPT | WT-CPT
Started | 42 | 40
Post-training Assessment | 31 | 32
Completed | 22 | 23
Not Completed | 20 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CEFT-CPT | WT-CPT | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.07 (8.14) | 38.40 (8.31) | 37.72 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 30 | 29 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 15 | 25
  Not Hispanic or Latino | 32 | 24 | 56
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 40 | 82
Education in years [Mean (Standard Deviation); unit: years] | 14.93 (1.83) | 15.25 (2.10) | 15.09 (1.96)

OUTCOME MEASURES:

1. Primary Outcome: Wisconsin Card Sorting Test (WCST)
Description: Wisconsin Card Sorting Test (WCST) is a neuropsychological measure of executive functioning, will be examined separately as well as in a composite with the other neuropsychological measures of executive functioning, range: -22 to 15, higher scores mean a worse outcome
Time Frame: change from baseline to completion of computerized cognitive training (6 weeks)
Population: Two participants did not complete this measure prior to being lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 29 | 32
score on a scale | -2.69 (4.24) | -1.47 (6.41)

2. Primary Outcome: Paced Auditory Serial Addition Test (PASAT)
Description: Paced Auditory Serial Addition Test (PASAT) is a neuropsychological measure of executive functioning, will be examined separately as well as in a composite with the other neuropsychological measures of executive functioning, range: -22 to 47, higher scores mean a better outcome
Time Frame: change from baseline to completion of computerized cognitive training (6 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 31 | 32
score on a scale | 14.32 (13.03) | 10.88 (14.61)

3. Primary Outcome: Delis Kaplan Executive Function System (D-KEFS)
Description: Delis Kaplan Executive Function System (D-KEFS) is a neuropsychological measure of executive functioning, will be examined separately as well as in a composite with the other neuropsychological measures of executive functioning, range: -39 to 27, higher scores mean a worse outcome
Time Frame: change from baseline to completion of computerized cognitive training (6 weeks)
Population: A participant was not able to complete this measure due to color blindness
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 31 | 31
score on a scale | -4.90 (8.83) | -3.81 (10.05)

4. Primary Outcome: Behavior Rating Inventory of Executive Function (BRIEF)
Description: Behavior Rating Inventory of Executive Function (BRIEF) is a self-report measure of executive functioning, items are summed to create a total score, range: -32 to 30, higher scores mean a worse outcome
Time Frame: change in subjective executive functioning from baseline to completion of computerized cognitive training (6 weeks)
Population: Two participants did not complete this measure prior to being lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 29 | 32
score on a scale | -6.52 (12.39) | -3.50 (16.29)

5. Primary Outcome: WAIS-IV Digit Span Sequencing Subtest
Description: Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) Digit Span Sequencing subtest is a neuropsychological measure of executive functioning, will be examined separately as well as in a composite with the other neuropsychological measures of executive functioning, range: -3 to 3, higher scores mean a better outcome
Time Frame: change from baseline to completion of computerized cognitive training (6 weeks)
Population: One participant did not complete this measure prior to being lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 30 | 32
score on a scale | 1.03 (1.63) | .31 (1.57)

6. Primary Outcome: N-Back Task Performance
Description: N-Back is a task that tests executive functioning, range: -.25 to .28, higher scores means a better outcome
Time Frame: change from baseline to completion of computerized cognitive training (6 weeks)
Population: Some participants were unable to complete this measure due to COVID restrictions related to in-person study visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 27 | 32
score on a scale | .04 (.12) | -.01 (.11)

7. Primary Outcome: Go/No-Go Task Performance
Description: Go/No-Go is a task that tests executive functioning, range: -.04 to .02, higher scores mean a worse outcome
Time Frame: change from baseline to completion of computerized cognitive training (6 weeks)
Population: Some participants were unable to complete this measure due to COVID restrictions related to in-person study visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 27 | 32
score on a scale | -.01 (.01) | -.001 (.02)

8. Secondary Outcome: Clinician-Administered PTSD Scale for DSM 5 (CAPS-5)
Description: Clinician-Administered PTSD Scale for DSM 5 (CAPS-5) is a clinical interview assessing PTSD symptoms that will be administered at 3 time points: baseline, after completion of cognitive training, and after completion of Cognitive Processing Therapy, range: -38 to 18, higher scores mean a worse outcome
Time Frame: change in PTSD symptoms from baseline to completion of Cognitive Processing Therapy (12 sessions completed after cognitive training), approximately 12 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 22 | 23
score on a scale | -8.18 (13.20) | -4.96 (11.67)

9. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: PTSD Checklist for DSM-5 (PCL-5) is a self-report questionnaire that will be administered at 15 time points: at baseline, after completion of cognitive training, at each of the 12 therapy sessions, and after completion of Cognitive Processing Therapy, range: -49 to 28, higher scores mean a worse outcome
Time Frame: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 22 | 23
score on a scale | -12.64 (17.85) | -11.70 (12.32)

10. Secondary Outcome: World Health Organization Quality of Life - BREF
Description: World Health Organization Quality of Life - BREF (WHOQOL-BREF) is a self-report questionnaire assessing quality of life that will be administered at 3 time points: baseline, after completion of cognitive training, and after completion of Cognitive Processing Therapy. Four subscales are computed (range 4-20): physical health, psychological, social relationships, and environment, range: -2.7 to 6.7, higher scores mean a better outcome
Time Frame: change in quality of life from baseline to completion of Cognitive Processing Therapy (12 sessions completed after cognitive training), approximately 12 weeks after baseline assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 22 | 23
score on a scale | 1.61 (2.52) | 1.39 (2.10)

11. Secondary Outcome: Time (in Minutes) Spent Completing Cognitive Processing Therapy Homework
Description: At each of the CPT sessions, participants will report how much time they spent completing homework since the previous session
Time Frame: time (in minutes) spent completing homework from CPT session 1 to CPT session 12 (across approximately 6 weeks, weeks 7-12 after baseline)
Population: Number of participants reflect only those participants who completed at least 2 sessions of CPT (i.e., enough sessions to complete at least one homework assignment)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 28 | 29
minutes | 426.68 (356.59) | 448.28 (610.06)

12. Secondary Outcome: Number of CPT Sessions Completed
Description: Number of CPT sessions completed out of a possible total of 12 sessions
Time Frame: CPT sessions completed (out of a possible 12) after completing the cognitive training (across approximately 6 weeks, weeks 7-12 after baseline)
Measure: Mean (Standard Deviation); unit: number of CPT sessions completed
Arm/Group | CEFT-CPT | WT-CPT
Number analyzed (Participants) | 42 | 40
number of CPT sessions completed | 6.76 (5.56) | 7.78 (5.31)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CEFT-CPT | WT-CPT
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03260127/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT03260127/ICF_001.pdf